CLINICAL TRIAL: NCT02228265
Title: Identifying Mechanisms of Resistance to Enzalutamide (MDV3100) Treatment in Men With Castration-Resistant Prostate Cancer
Brief Title: Molecular Features and Pathways in Predicting Drug Resistance in Patients With Metastatic Castration-Resistant Prostate Cancer Receiving Enzalutamide
Status: Completed | Type: Observational
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Tom Beer, Principal Investigator, OHSU Knight Cancer Institute
Other Study IDs: IRB00009259; NCI-2014-01438 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MR00046920; IRB00009259 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2014-08-25; First posted 2014-08-29 (Estimated); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Castration Levels of Testosterone; Castration-Resistant Prostate Carcinoma; Prostate Adenocarcinoma; PSA Progression; Recurrent Prostate Carcinoma; Stage IV Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzalutamide

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue and blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Ancillary-Correlative (genetic analysis): Patients undergo collection of blood and tissue samples at baseline, during administration of enzalutamide and after the time of disease progression for analysis via immunohistochemistry, comparative genome hybridization, and sequencing.
  Interventions: Other: Cytology Specimen Collection Procedure; Drug: Enzalutamide; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Other: Cytology Specimen Collection Procedure — Undergo blood and tissue collection
  Other Names: Cytologic Sampling
Drug: Enzalutamide — Given PO
  Other Names: ASP9785; MDV3100; Xtandi
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This research trial studies molecular features and pathways in predicting drug resistance in patients with castration-resistant prostate cancer that has spread to other parts of the body and who are receiving enzalutamide. Studying samples of blood and tissue in the laboratory from patients receiving enzalutamide may help doctors learn more about molecular features and pathways that may cause prostate cancer to be resistant to the drug.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the correlations between baseline molecular features and pathways and prostate-specific antigen (PSA) response (</>= 50% decline) at 12 weeks versus (vs.) baseline.

SECONDARY OBJECTIVES:

I. To assess the correlations between the baseline molecular features and pathways and progression-free survival (defined as time from day 1 of study drug treatment to date of radiographic progression or clinical progression), disease-specific survival (defined as the time from day 1 of study drug to date of death from prostate cancer), and overall survival (defined as time from day 1 of study drug treatment to date of death from any cause).

II. To assess the correlations between the baseline molecular features and pathways and time to PSA progression.

III. To identify molecular features and cellular pathways present in tumors from men with metastatic castrate-resistant prostate cancer (CRPC) that are progressing despite enzalutamide treatment.

IV. To explore correlation between baseline molecular features and pathways and objective response.

V. To assess the correlations between the baseline molecular features and pathways and degree of PSA decline at 12 weeks and maximal PSA decline observed while on study.

VI. To assess the correlations between the baseline molecular features and time on treatment.

TERTIARY OBJECTIVES:

I. To assess correlations between cell-free deoxyribonucleic acid (cfDNA) molecular features from blood and molecular features and pathways from the biopsy samples.

II. To assess correlations between cfDNA molecular features and endpoints in the primary and secondary objectives listed above.

III. To explore correlations with baseline molecular features and tissue histology.

IV. To explore correlations with baseline tissue histology and PSA change, time to PSA progression, time on treatment, progression-free survival, and overall survival.

OUTLINE:

Patients undergo collection of blood and tissue samples at baseline, during administration of enzalutamide, and after the time of disease progression for analysis via immunohistochemistry, comparative genome hybridization, and sequencing.

After completion of study, patients are followed up every 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate without neuroendocrine differentiation or small cell features
* Ongoing androgen deprivation therapy with a gonadotropin-releasing hormone (GnRH) analogue or orchiectomy (i.e., surgical or medical castration); for patients who have not had an orchiectomy, there must be a plan to maintain effective GnRH-analogue therapy for the duration of the trial
* Radiographic evidence of regional or distant metastases with suspected tumor in an area that is safe to biopsy
* Willingness to undergo a tumor biopsy at baseline and at disease progression
* Serum testosterone level < 50 ng/dL at screening
* Progressive disease by PSA or imaging in the setting of medical or surgical castration; disease progression for study entry is defined as one or more of the following three criteria:

  * PSA progression defined by a minimum of three rising PSA levels with an interval of >= 1 week between each determination; the PSA value at screening should be >= 2 ug/L (2 ng/ml)
  * Soft tissue disease progression defined by Response Evaluation Criteria in Solid Tumors (RECIST 1.1)
  * Bone disease progression defined by two or more new lesions on bone scan
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Clinically able, in the opinion of the investigator, to receive MDV3100 (enzalutamide)
* Willing and able to give informed consent
* A minimum of 4 weeks elapsed off of anti-androgen therapy prior to enrollment for flutamide and 6 weeks for bicalutamide and nilutamide without evidence of an anti-androgen withdrawal response; patients who NEVER HAD A PSA decline with the most recent anti-androgen therapy or in whom the response to the most recent anti-androgen was for < 3 months require only a 2 week washout period prior to first dose of study drug

Exclusion Criteria:

* Severe, concurrent disease, infection, or co-morbidity that, in the judgment of the investigator, would make the patient inappropriate for enrollment
* Metastases in the brain or active epidural disease (NOTE: patients with treated epidural disease are allowed)
* Platelet count < 75,000/uL
* Prothrombin time (PT) or international normalized ratio (INR) and a partial thromboplastin time PTT > 1.5 times the institutional upper limit of normal (ULN)
* Structurally unstable bone lesions suggesting impending fracture
* Previous treatment with MDV3100, ARN-509, or BMS-641988
* Medical contraindications to stopping aspirin, Coumadin or other anticoagulants for 1 week prior to image-guided tumor biopsies
* Plans to initiate treatment with an investigational agent while on study prior to discontinuation of MDV3100 treatment
* A second active malignancy except adequately treated non-melanoma skin cancer or other non-invasive or in situ neoplasm

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with prostate cancer treated at Oregon Health and Science University Knight Cancer Institute
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2013-03-12 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2020-02-27 (Actual)

PRIMARY OUTCOMES:
PSA response, a binary variable indicating whether the PSA level has declined >= 50% within 12 weeks of beginning enzalutamide treatment | Within 12 weeks
  Will be reported with 95% exact confidence interval.

SECONDARY OUTCOMES:
Degree of PSA decline | 12 weeks
  Simple linear regression will be used to assess the association between molecular biomarker predictors and the continuous endpoints. Logarithm transformation or other forms of transformation may be conducted to the continuous endpoints to address the skewedness of the distributions if necessary.
Disease-specific survival | Time from day 1 of the study drug to date of death from prostate cancer, assessed up to 4 years
  Will be graphically illustrated using Kaplan-Meier plots of estimated survival distribution for patients (</>= 50%) PSA decline at 12 weeks. Log-rank test will be fitted to determine whether the estimated survival distribution of each time-to-event endpoint differs for patients with PSA decline >= 50% versus patients with PSA decline < 50%. Cox regression models will be fitted to obtain the estimated hazard ratio for each time-to-event endpoints for patients who had >= 50% PSA decline at 12 weeks versus those who had not.
Maximal PSA decline observed while on study | Up to 4 years
  Simple linear regression will be used to assess the association between molecular biomarker predictors and the continuous endpoints. Logarithm transformation or other forms of transformation may be conducted to the continuous endpoints to address the skewedness of the distributions if necessary.
Molecular features | Up to 4 years
  Will assess correlations between the baseline molecular features and time on treatment.
Objective response | Up to 4 years
  Will be summarized using the estimated proportion and 95% confidence interval. Simple logistic regression model will be used to assess the association between molecular biomarker predictors and these binary secondary endpoints.
Overall survival | Time from day 1 of study drug treatment to date of death from any cause, assessed up to 4 years
  Will be graphically illustrated using Kaplan-Meier plots of estimated survival distribution for patients (</>= 50%) PSA decline at 12 weeks. Log-rank test will be fitted to determine whether the estimated survival distribution of each time-to-event endpoint differs for patients with PSA decline >= 50% versus patients with PSA decline < 50%. Cox regression models will be fitted to obtain the estimated hazard ratio for each time-to-event endpoints for patients who had >= 50% PSA decline at 12 weeks versus those who had not.
Progression for a subgroup of patients who have metastatic castration resistant prostate cancer and have received enzalutamide treatment | Up to 4 years
  Will be summarized using the estimated proportion and 95% confidence interval. Simple logistic regression model will be used to assess the association between molecular biomarker predictors and these binary secondary endpoints.
Progression-free survival | Time from day 1 of study drug treatment to date of first documented radiographic progression or clinical progression, assessed up to 4 years
  Will be graphically illustrated using Kaplan-Meier plots of estimated survival distribution for patients (</>= 50%) PSA decline at 12 weeks. Log-rank test will be fitted to determine whether the estimated survival distribution of each time-to-event endpoint differs for patients with PSA decline >= 50% versus patients with PSA decline < 50%. Cox regression models will be fitted to obtain the estimated hazard ratio for each time-to-event endpoints for patients who had >= 50% PSA decline at 12 weeks versus those who had not.
Time to PSA progression | Up to 4 years
  Will be graphically illustrated using Kaplan-Meier plots of estimated survival distribution for patients (</>= 50%) PSA decline at 12 weeks. Log-rank test will be fitted to determine whether the estimated survival distribution of each time-to-event endpoint differs for patients with PSA decline >= 50% versus patients with PSA decline < 50%. Cox regression models will be fitted to obtain the estimated hazard ratio for each time-to-event endpoints for patients who had >= 50% PSA decline at 12 weeks versus those who had not.

CONTACTS AND LOCATIONS:
Overall Officials: Joshi Alumkal, Principal Investigator — OHSU Knight Cancer Institute
Locations (3):
- United States (3):
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - OHSU Knight Cancer Institute, Portland, Oregon